CLINICAL TRIAL: NCT05325736
Title: Improvement in Glycemic Response After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Weizmann Institute of Science (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0046-21-TLV
Record Dates: First submitted 2022-02-10; First posted 2022-04-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool, serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- sleeve gastrectomy surgery: participants undergoing sleeve gastrectomy surgery for weight reduction
  Interventions: Procedure: sleeve gastrectomy surgery
- gastric bypass surgery: participants undergoing gastric bypass surgery for weight reduction
  Interventions: Procedure: gastric bypass surgery
- cholecystectomy: participants undergoing cholecystectomy
  Interventions: Procedure: control
- Pancreatectomy: participants undergoing Pancreatectomy
  Interventions: Procedure: Pancreatectomy

INTERVENTIONS:
Procedure: sleeve gastrectomy surgery — participants undergoing sleeve gastrectomy surgery
  Groups: sleeve gastrectomy surgery
Procedure: gastric bypass surgery — participants undergoing gastric bypass surgery
  Groups: gastric bypass surgery
Procedure: control — cholecystectomy
  Groups: cholecystectomy
Procedure: Pancreatectomy — Collecting a sample of an unidentified healthy pancreas to extract insulin-secreting beta cells from the sample
  Groups: Pancreatectomy

SUMMARY:
decipher the role of microbiota in glycemic response change after bariatric surgery

DETAILED DESCRIPTION:
Despite the vast knowledge linking the gut microbiome to metabolism and the glucose response, the relation still remains unclear. hopefully, a deep understanding of the mechanisms underlying metabolic improvement following bariatric surgery will make it possible to identify targets for pharmacological intervention, which will reduce the need for surgery and its risks.

Previous studies have characterized the microbiome after bariatric surgery, but most suffer from methodological limitations.

The current study has the potential to be innovative and make a significant contribution to understanding the mechanisms involved in early metabolic improvement after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* candidates of bariatric surgery or cholecystectomy
* age 18-70
* male/female

Exclusion Criteria:

* previous bariatric surgery
* type 1 diabetes
* antibiotic treatment 3 months prior to the study
* probiotic treatment 3 months prior to the study
* chronic disease - gastrointestinal disease, malignancy, psychiatric disorder, endocrinologic disorders
* any pathologic findings during endoscopy
* participants who will suffer from a post-operation complication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients arriving at the outpatient unit at Tel Aviv Sourasky medical center
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic response | up to 4 years
  The glycemic response will be measured by taking a blood test (glucose) after 12 hours fast and a second blood test (glucose) after an OGTT(oral glucose tolerance test) of 50 g glucose
microbiota composition | up to 4 years
  The microbiota composition will be assessed using the stool samples of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Avner Leshem, MD, Study Director — Weizmann institute; Danit Dayan, MD, Principal Investigator — Souraski medical center
Locations (2):
- Israel (2):
  - Weizmann Institute of Science, Rehovot
  - Souraski medical center, Tel Aviv